CLINICAL TRIAL: NCT03340012
Title: Clinical and Radiographic Evaluation of Guided Tissue Regeneration With Radiation-sterilized Allogenic Bone Grafts or Xenogenic Grafts for the Treatment of Intrabony Defects in Aggressive Periodontitis: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Guided Tissue Regeneration With Radiation-sterilized Allogenic Bone Grafts or Xenogenic Grafts for the Treatment of Intrabony Defects in Aggressive Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WUM.PERIO.02
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Periodontitis, Aggressive
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GTR + radiation-sterilize allogenic bone graft (TEST) (Experimental): The surgical procedure will be performed in line with minimally invasive surgical technique by Cortellini and Tonetti (2007). The intrabony defects will be debrided and the roots will be planned. The required quantity of radiation-sterilized allogenic bone graft will be delivered into intrabony defects. Subsequently, a trimmed collagen membrane will be placed over graft. The flaps will be sutured with non-absorbable modified internal mattress sutures.
  Interventions: Device: GTR + radiation-sterilize allogenic bone graft
- GTR + xenogenic graft (CONTROL) (Active Comparator): The surgical procedure will be performed in line with minimally invasive surgical technique by Cortellini and Tonetti (2007). The intrabony defects will be debrided and the roots will be planned. The required quantity of xenogenic graft will be delivered into intrabony defects. Subsequently, a trimmed collagen membrane will be placed over graft. The flaps will be sutured with non-absorbable modified internal mattress sutures.
  Interventions: Device: GTR + xenogenic graft

INTERVENTIONS:
Device: GTR + radiation-sterilize allogenic bone graft — Guided tissue regeneration of intrabony defects with collagen membrane (Bio-Gide® Perio, Geistlich Biomaterials) and radiation-sterilized allogenic bone graft from the Central Tissue Bank in Warsaw
  Arms: GTR + radiation-sterilize allogenic bone graft (TEST)
Device: GTR + xenogenic graft — Guided tissue regeneration of intrabony defects with collagen membrane (Bio-Gide® Perio, Geistlich Biomaterials) and xenogenic graft (Bio-Oss®, Geistlich Biomaterials)
  Arms: GTR + xenogenic graft (CONTROL)

SUMMARY:
The treatment of intrabony defects in patients with aggressive periodontitis remains a challenging procedure and novel therapeutic strategies are sought. The purpose of this study is to compare the clinical and radiographic outcomes of using guided tissue regeneration (GTR) with radiation-sterilized allogenic bone grafts (material prepared in the Central Tissue Bank in Warsaw, Poland) versus guided tissue regeneration with xenogenic grafts (Bio-Oss®, Geistlich Biomaterials, Princeton, New Jersey, United States) in the treatment of localized intrabony defects in patients with aggressive periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of aggressive periodontitis in line with American Academy of Periodontology classification (Lang et al. 1999)
* Familial aggregation (history of periodontitis in parents or siblings)
* Presence of at least two teeth with probing pocket depth (PPD) ≥ 6mm and clinical attachment level (CAL) ≥ 5 mm associated with an intrabony defect of at least 3 mm as detected in diagnostic periapical radiographs
* No furcation involvement of the teeth presenting the intraosseous defects
* The width of keratinized tissue on the facial aspect of the selected teeth ≥ 2 mm

Exclusion Criteria:

* Full-mouth plaque index ≥ 20% (Ainamo & Bay 1975)
* Full-mouth sulcus bleeding index ≥ 15% (Mühlemann & Son 1971)
* Smoking more than 10 cigarettes/day
* Systemic diseases with compromised healing potential of infectious diseases
* Drugs affecting periodontal health / healing
* Pregnant and lactating females
* Previous periodontal surgery in the area

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-05 (Estimated); Primary Completion 2019-05-05 (Estimated); Study Completion 2019-05-05 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical attachment level (CAL) | Baseline and 12 months after surgery
  CAL will be measured in millimeters on the study teeth at 6 locations as a distance from the cementoenamel junction to the bottom of the gingival sulcus. The average differences between 12 months and baseline measurements at the sites with the most advanced attachment loss at baseline will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw, Warsaw, Mazowsze, Poland